CLINICAL TRIAL: NCT06414083
Title: Histologic Comparison of Ablative Techniques for Endometriosis - a Randomized Trial
Brief Title: Histologic Comparison of Ablative Techniques for Endometriosis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: TriHealth Inc. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 24-007
Record Dates: First submitted 2024-05-10; First posted 2024-05-16 (Actual); Last update posted 2024-05-30 (Actual); Status verified 2024-05

CONDITIONS: Endometriosis; Endometriosis-related Pain; Endometriosis Pelvic; Endometriosis; Peritoneum
MeSH Terms: conditions — Endometriosis | interventions — Diathermy; Lasers, Gas

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Pathologist is blinded to treatment arm
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (3):
- Diathermy (Active Comparator)
  Interventions: Device: Diathermy
- CO2 Laser (Active Comparator)
  Interventions: Device: CO2 Laser
- Argon Beam Coagulator (Active Comparator)
  Interventions: Device: Argon Beam Coagulator

INTERVENTIONS:
Device: Diathermy — Diathermy will be used to ablate the randomized sample.
  Arms: Diathermy
Device: CO2 Laser — CO2 Laser will be used to ablate the randomized sample.
  Arms: CO2 Laser
Device: Argon Beam Coagulator — Argon Beam Coagulator will be used to ablate the randomized sample.
  Arms: Argon Beam Coagulator

SUMMARY:
To our knowledge, no other human studies directly compare the effectiveness of the various ablative technologies. We set out to design a study to directly compare ablative energy sources and evaluate their ability to destroy native endometriosis tissue in humans.

ELIGIBILITY:
Inclusion Criteria:

* Adult women 18 years of age or older
* Already planning to undergo scheduled robotic assisted or laparoscopic excision of lesions for pelvic pain symptoms (pelvic pain, dysmenorrhea, dyspareunia, dysuria, dyschezia, ovarian pain) or endometriosis of any kind (endometriosis of any location, or endometrioma)

Exclusion Criteria:

* Known pregnancy at enrollment or at the time of the excision surgery

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 141 (Estimated)
Dates: Start 2024-05-09 (Actual); Primary Completion 2025-05-09 (Estimated); Study Completion 2025-06-09 (Estimated)

PRIMARY OUTCOMES:
Positive Histology | 0 days
  Endometriosis seen on pathologic sample.

SECONDARY OUTCOMES:
Pelvic Pain | 3 months
  Pre-operative and Post-operative Pelvic Pain Visual Analog Scale. Minimum Score 0. Maximum Score 100. Higher score is worse outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- Good Samaritan Hospital, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Namaky DD, Carrel-Lammert M, Hoehn J, Yeung J. Histologic Comparison of Ablative Techniques for Endometriosis: a Randomized Trial. J Minim Invasive Gynecol. 2026 Jan 10:S1553-4650(26)00044-0. doi: 10.1016/j.jmig.2026.01.020. Online ahead of print. PMID 41525928